CLINICAL TRIAL: NCT07104188
Title: Effects of Energy Drink on Repeated Sprint Performance and Cognitive Function in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chien-Wen Hou (Other)
Responsible Party: Sponsor-Investigator, Chien-Wen Hou, professor, University of Taipei
Organization: University of Taipei (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-2021-021
Record Dates: First submitted 2025-07-01; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2022-06

CONDITIONS: Exercise Performance Impairment; Cognitive Function Decline; Fatigue
Keywords: sports supplements; Caffeine; anserine; elderberry; high-intensity exercise
MeSH Terms: conditions — Fatigue | interventions — Caffeine; Energy Drinks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group (Placebo Comparator): Participants in this group received a placebo supplement that contained no active ingredients.
  Interventions: Dietary Supplement: A non-active placebo supplement.
- Caffeine Group (Active Comparator): Participants in this group received a caffeine supplement containing 220 mg of caffeine.
  Interventions: Dietary Supplement: Caffeine
- Energy Drink Group (Experimental): Participants in this group received an energy drink containing 220 mg of caffeine, 1800 mg of anserine extract, and 400 mg of elderberry extract.
  Interventions: Dietary Supplement: Energy Drink

INTERVENTIONS:
Dietary Supplement: A non-active placebo supplement. — Placebo powder mixed into 100 ml grape juice and 200 ml water, consumed 30 minutes before testing.
  Arms: Placebo Group
Dietary Supplement: Caffeine — 220 mg caffeine powder mixed into 100 ml grape juice and 200 ml water, consumed 30 minutes before testing.
  Arms: Caffeine Group
Dietary Supplement: Energy Drink — A supplement containing 220 mg caffeine, 1800 mg anserine extract, and 400 mg elderberry extract, mixed into 100 ml grape juice and 200 ml water, consumed 30 minutes before testing.
  Arms: Energy Drink Group

SUMMARY:
Energy drinks are often used by athletes before competitions to enhance their performance. Recent research has pointed out that the performance effects of select ingredients have been studied individually but not in combination with caffeine. Therefore, this study is designed to investigate the effects of caffeine, anserine, and elderberry on cognitive function and repeated sprint performance of athletes during a high-intensity exercise protocol.

A double-blind, randomized crossover design will be employed. Three types of supplements will be tested: placebo, caffeine (220 mg), and an energy drink containing 220 mg caffeine, 288 mg anserine, 400 mg elderberry, and 660 mg of a vitamin-mineral mixture. Twelve college athletes will be recruited to complete repeated sprint tests on a cycle ergometer until exhaustion and to undertake a series of cognitive tasks during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-25
* Currently enrolled college student
* Active members of a collegiate wrestling team (college wrestlers)
* Engaged in regular wrestling training
* Willing and able to provide written informed consent
* Agreed to maintain their usual diet and training frequency during the study period

Exclusion Criteria:

* Individuals with known caffeine sensitivity
* Any existing health condition that may interfere with high-intensity exercise (e.g., cardiovascular, metabolic, or neurological disorders)
* Inability or unwillingness to follow study instructions

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Repeated Sprint Performance | From second to fourth weeks, 30 minutes after the participants consumed the supplement.
  Participants completed a repeated sprint test on a cycle ergometer after supplement intake and 30 minutes waiting. The test involved multiple 10-second maximal sprints with 20-second passive recoveries, continuing until fatigue (cadence < 70 rpm for over 3 seconds). During the test, the resistance was set at 0.8 Nm/kg body weight. Total power output during repeated sprint performance was the primary outcome.

SECONDARY OUTCOMES:
Squares performance- spatial working memory | From the fifth -seventh weeks, 30 minutes after the participants consumed the supplement.
  The spatial memory task required participants to recall the spatial location of dots presented on a screen. A 6×6 grid was shown. First, some squares were colored for one second, and after they re-turned to normal, we need to press the squares that were previously colored. It would end if participants answered incorrectly. At higher stages, more squares were randomly colored. Reaching higher stages indicates better memory performance.
Colour drop performance- executive function | From the fifth -seventh weeks, 30 minutes after the participants consumed the supplement.
  evaluates executive function by asking participants to name the ink color of color-words that are incongruent (e.g., the word "GREEN" printed in blue ink). Incorrect responses end the test; higher scores indicate better executive function.
Schulte grid performance- attention | From the fifth -seventh weeks, 30 minutes after the participants consumed the supplement.
  Schulte Grid Test - measures attention by requiring participants to find numbers from 1 to 36 in ascending order on a 6×6 grid as quickly as possible; faster completion indicates better attention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Taipei, Taipei, Taiwan